CLINICAL TRIAL: NCT03740308
Title: Evaluating the Performance and Efficiency of Zirconia Crowns in Treating Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Pedo-01-2018
Record Dates: First submitted 2018-08-24; First posted 2018-11-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Primary Teeth
Keywords: Primary posterior teeth; zirconia crown

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinded study (Patients blinding & Outcome-assessor blinding).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locally Made Zirconia Crowns (Active Comparator): One operator completes all the teeth preparing and restoring procedures. Local anesthesia is achieved using Lidocaine Hydrochloride 2% with Epinephrine 1:100,000. The teeth are then isolated using a rubber dam. After caries excavation, the teeth are prepared according to manufacturer instructions.
  Interventions: Device: Locally Made Zirconia Crowns
- ZR Zirconia Crwons NuSmile ® Crowns (Experimental): One operator completes all the teeth preparing and restoring procedures. Local anesthesia is achieved using Lidocaine Hydrochloride 2% with Epinephrine 1:100,000. The teeth are then isolated using a rubber dam. After caries excavation, the teeth are prepared according to manufacturer instructions. (Same as Arm 1 Description)
  Interventions: Device: ZR Zirconia Crwons NuSmile ® Crowns

INTERVENTIONS:
Device: Locally Made Zirconia Crowns — Occlusal reduction by decreasing the occlusal surface to less than the natural occlusal profile by about 1-1.5 mm roughly. Proximal reduction by unfastening the interproximal contacts. The tooth should be trimmed down circumferentially by around 0.5-1.25 mm as needed. Subgingival reduction, leaving no undercuts or subgingival ridges, about 1-2 mm subgingivally on every area should be prepared. Completion of the preparation by eliminating sharp lines and pointed angles to allow all prepared areas to be marginally rounded and smoothed. Locally Made Zirconia Crowns are fixed using Glass Ionomer cement (Fuji- Jaban).
  Arms: Locally Made Zirconia Crowns
Device: ZR Zirconia Crwons NuSmile ® Crowns — Occlusal reduction by decreasing the occlusal surface to less than the natural occlusal profile by about 1-1.5 mm roughly. Proximal reduction by unfastening the interproximal contacts. The tooth should be trimmed down circumferentially by around 0.5-1.25 mm as needed. Subgingival reduction, leaving no undercuts or subgingival ridges, about 1-2 mm subgingivally on every area should be prepared. Completion of the preparation by eliminating sharp lines and pointed angles to allow all prepared areas to be marginally rounded and smoothed. ZR Zirconia Crwons NuSmile ® Crowns are fixed using Glass Ionomer cement (Fuji- Jaban).
  Arms: ZR Zirconia Crwons NuSmile ® Crowns

SUMMARY:
This randomized clinical trial aims to compare the clinical outcomes of two full-coronal-coverage restorations (locally-made preformed Zirconia crowns [LMP] and NuSmile Zirconia crowns [Nu/ZR]) in treating carious primary teeth. Amongst the children attending the clinics of the Dental School at Damascus University, the ones having an indication for crowns restorations will be screened and if they are conformant to the inclusion criteria then they will be recruited until 60 teeth are reached (30 teeth for LMP/ZR restorations and 30 for Nu/ZR restorations).

DETAILED DESCRIPTION:
This randomized clinical trial compares the clinical outcomes of using two full-coronal zirconia restorations (locally-made preformed zirconia crowns, and NuSmile zirconia crowns) in treating carious primary teeth. Children attending to the clinics of the Faculty of Dentistry - Damascus University and who happen to be in need for dental restorations will be screened for the study's inclusion criteria till 60 teeth are recruited (30 teeth for locally made preformed zirconia crowns restorations and 30 for NuSmile zirconia crowns restorations). One crown only will be used for each patient (totally 60 patients) to ensure equalizing the variables for both groups. The randomization will be done using SPSS software version 20.0 (Armonk, NY; IBM Corp., USA). The study is going to be a double-blinded study (Patients blinding and Outcomes-assessor blinding). Simple descriptive statistics will be used for the analysis, also using Wilcoxon Signed-Rank test. The level of significance will be set at (α = 0.05) and the level of confidence at (95%). The intervention is preparing primary molars which have one or more indications for crowning, and according to manufacturer instructions. Then following up the treated primary molars for 1 month, 3 months, and 6 months intervals. The main goals are measuring and comparing the status of the gingiva and any improvements in the gingival health relative to the intervention, the plaque retention in regard to the gingival response to the material of restoration, and also the crowns resistance to changes, despite its high cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the age group of 4 to 8 years of age.
* Patients with good oral hygiene.
* Healthy children, i.e. free of any systematic diseases or any developmental disturbances of the teeth and jaws
* A minimal of two surfaces of caries in the targeted tooth
* Corresponding treated teeth has not got any crown earlier
* Patients with ECC as defined by the American Academy for Pediatric Dentistry.
* Cooperative patients who have a dental behavioral assessment of "definitely positive" according to Frankl behavior classification scale.

Exclusion Criteria:

* No patient is excluded by gender, race, or due to socio-economic backgrounds.

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Changes of crowns integrity | Evaluating after 1 month, 3 months, 6 months
  Crowns integrity changes will be measured with the naked eye and the light cure device. The scores are as follows: (0 = No crack, No fracture, No chip) (1 = Chip) (2 = Crack) (3 = Fracture). (Cvar and Rygp 2005)

SECONDARY OUTCOMES:
Changes of gingival index | Evaluating after 1 month, 3 months, 6 months
  is measured by passing the periodontal probe tip gently within the sulcus around each crowned tooth. The scores are as follows: (0 = normal gingiva) (1= mild inflammation) (2 = Moderate inflammation) (3 = severe inflammation). (Loe and Silness 1963)
Changes of crown marginal adaptation | Evaluating after 1 month, 3 months, 6 months
  Crown marginal adaptation will be measured at the buccal and lingual walls and will be referred to as either good for crowns with sealed margins or poor when the explorer detects an open margin. (Farsi and Sharaf 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AlTinawi, PhD., Study Director — Professor - Pediatric Dentistry Department - Faculty of Dentistry - Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Pedodontics, Damascus University

REFERENCES:
- [Result] Aiem E, Smail-Faugeron V, Muller-Bolla M. Aesthetic preformed paediatric crowns: systematic review. Int J Paediatr Dent. 2017 Jul;27(4):273-282. doi: 10.1111/ipd.12260. Epub 2016 Aug 17. PMID 27532506
- [Result] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Result] Fuks AB, Ram D, Eidelman E. Clinical performance of esthetic posterior crowns in primary molars: a pilot study. Pediatr Dent. 1999 Nov-Dec;21(7):445-8. PMID 10633519
- [Result] Sharaf AA, Farsi NM. A clinical and radiographic evaluation of stainless steel crowns for primary molars. J Dent. 2004 Jan;32(1):27-33. doi: 10.1016/s0300-5712(03)00136-2. PMID 14659715
- [Result] Mittal HC, Goyal A, Gauba K, Kapur A. Clinical Performance of Indirect Composite Onlays as Esthetic Alternative to Stainless Steel Crowns for Rehabilitation of a Large Carious Primary Molar. J Clin Pediatr Dent. 2016;40(5):345-52. doi: 10.17796/1053-4628-40.5.345. PMID 27617373
- [Result] Croll TP, Helpin ML. Preformed resin-veneered stainless steel crowns for restoration of primary incisors. Quintessence Int. 1996 May;27(5):309-13. PMID 8941812
- [Result] Shah PV, Lee JY, Wright JT. Clinical success and parental satisfaction with anterior preveneered primary stainless steel crowns. Pediatr Dent. 2004 Sep-Oct;26(5):391-5. PMID 15460292